CLINICAL TRIAL: NCT02945592
Title: Active Cue-Training in Neglect
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Klinikum Bremen Ost (Other)
Responsible Party: Principal Investigator, Nergiz Turgut, MSc, Klinikum Bremen Ost
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 367915
Record Dates: First submitted 2016-10-19; First posted 2016-10-26 (Estimated); Last update posted 2018-03-06 (Actual); Status verified 2018-03

CONDITIONS: Hemispatial Neglect
Keywords: Hemispatial Neglect; cueing; egocentric-allocentric; early rehabilitation; parietal tDCS
MeSH Terms: conditions — Perceptual Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): * adaptive, therapeutic cueing during reading tasks
  * adaptive, therapeutic cueing during visuo spatial tasks
  Interventions: Behavioral: Cueing
- Control (No Intervention): - unspecific neglect treatment

INTERVENTIONS:
Behavioral: Cueing
  Arms: Intervention

SUMMARY:
The presented study investigates standardized visual cueing in reading and visual spatial task as a treatment method for spatial neglect. In a randomized controlled design patients receive either cued reading and visual spatial tasks (intervention) or treatment which is unspecific to neglect (control).

In the intervention condition, patients with left-sided neglect receive intense training, including reading and visual spatial task with standardized and adapted visual cueing by the therapist. Improvements in reading and visual spatial tasks lead to a reduction of cues by the therapist. Accordingly, the patient has to apply self-cueing over time in order to solve the task.

For the control condition, all patients receive unspecific treatment without any standardized adapted cueing implemented by the therapist.

To enhance the effectivity of cueing in reading and visual spatial tasks, the investigators additionally conduct parietal transcranial direct current stimulation (tDCS) in those patients without tDCS exclusion criteria (see exclusion criteria below).

It is hypothesised that systematic and adaptive therapeutic cueing leads to a significant reduction of omissions of word and word parts in reading.

UPDATE: No Add-on tDCS was performed since it was not applicable for our severly impaired patients due to the strict exclusion criteria of tDCS.

ELIGIBILITY:
Inclusion Criteria:

* Left sided neglect
* Capacity of at least 30 minutes
* Ability to read in German language
* Mobilization of 80%

Exclusion Criteria:

* Previous known dementia
* Normal pressure hydrocephalus

Exclusion Criteria for tDCS Add-on (not exclusion of the intervention):

* Shunt
* Craniectomy
* Epilepsy
* Other metal implants

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2016-10; Primary Completion 2017-11 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Change in word and word-part omissions in standardized reading of text and word list | Primary Outcome Measure is assessed two times in the first week (3 days in between), after week 4, after week 7, after week 8
  the patient has to read a standardized text of 55 words and a word list of 13 words. Omissions of the complete word and/or of a word part are counted.

SECONDARY OUTCOMES:
Change in standardized evaluation of the body posture | Secondary Outcome Measure is assessed two times in the first week (3 days in between), after week 4, after week 7, after week 8
  A blinded neurologist evaluates spontaneous and cued body posture (head, eyes, trunk) for ipsilesional, moderate ipsilesional or no deviation.
Change in Apples Cancellation Task | Secondary Outcome Measure is assessed two times in the first week (3 days in between), after week 4, after week 7, after week 8
  a standardized measurement for the evaluation of egocentric and allocentric neglect symptoms
Change in activities of daily living using the Catherine Bergego Scale | Secondary Outcome Measure is assessed after week 1, after week 4, after week 7, after week 8
  The blinded hospital staff evaluates activities of daily living by using the Catherine Bergego scale with specified scoring criteria

CONTACTS AND LOCATIONS:
Overall Officials: Helmut Hildebrandt, Prof. Dr., Study Director — Universität Oldenburg, Klinikum Bremen-Ost
Locations (1):
- Klinikum Bremen-Ost, Bremen, Germany

IPD SHARING:
Plan to Share IPD: Undecided